CLINICAL TRIAL: NCT04305769
Title: Alanyl-glutamine Supplementation of Standard Treatment for C. Difficile Infection: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Alanyl-glutamine Supplementation for C. Difficile Treatment (ACT)
Acronym: ACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Carilion Clinic (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Cirle Warren, MD, Research Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200046
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Clostridioides Difficile Infection; Clostridium Difficile Infection; Clostridium Difficile Diarrhea; Clostridia Difficile Colitis
MeSH Terms: conditions — Clostridium Infections; Enterocolitis, Pseudomembranous | interventions — alanylglutamine; Glutamine

STUDY DESIGN:
Intervention Model Description: Block randomization will be applied to assign participants to one of the four study groups, either one of the three experimental (AQ) or control (placebo) group in 1:1:1:1 allocation from a list containing the randomized and blinded treatment assignments.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Alanyl-glutamine 0g (Placebo Comparator)
  Interventions: Drug: Alanyl-glutamine
- Alanyl-glutamine 4g (Experimental)
  Interventions: Drug: Alanyl-glutamine
- Alanyl-glutamine 24g (Experimental)
  Interventions: Drug: Alanyl-glutamine
- Alanyl-glutamine 44g (Experimental)
  Interventions: Drug: Alanyl-glutamine

INTERVENTIONS:
Drug: Alanyl-glutamine — The study agent is AQ, a dipeptide with a glutamine amino group joined to an alanyl residue. It has the following chemical structure: C8H15N3O4. It is a non-animal product available in the form of white crystals or crystalline powder. It is odorless, tasteless, stable and highly soluble.
  Other Names: Alagln; AQ; glutamine

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to determine the optimal dose and safety of oral alanyl-glutamine between 4, 24, and 44 g doses administered for 10 days with standard therapy among first time incident cases of uncomplicated C. difficile infection (CDI) in hospitalized, or outpatient, persons aged 18 or older. The investigators hypothesis is that alanyl-glutamine supplementation will decrease recurrence and mortality from CDI and these outcomes will be associated with improvement of inflammatory markers and restoration of intestinal microbiota function.

DETAILED DESCRIPTION:
This is a Phase II randomized, placebo-controlled, double-blinded, dose-ranging study to determine optimal effective dose and safety of AQ between 0, 4, 24, and 44 g doses administered orally for ten days concurrent with standard treatment (oral vancomycin or fidaxomicin at UVa) among cases of CDI in hospitalized persons, persons who are referred to the UVA C. difficile clinic or Carilion Hospital, age 18 and older. The investigators hypothesis is that AQ will reduce recurrence (primary outcome) and mortality (secondary outcome) at 60 days post-treatment. Furthermore, the investigators hypothesize that alanyl-glutamine supplementation will be associated with decreased intestinal and systemic inflammation and improvement of intestinal microbial and metabolic profiles. The investigators plan to enroll 260 patients, equally divided into 4 arms. Upon enrollment, participants will be randomized to either receive AQ at 4, 24, or 44 g or placebo (water). Study agent is administered once a day, orally or enterally, if feeding tube is present. Because the investigators are enrolling subjects over a longer period of time, block randomization will be used to ensure that relative temporal balance is maintained throughout the trial. Participants will be followed up daily during treatment for adverse event monitoring and weekly for 60 days post-treatment for recurrences and survival. Blood, urine and stool specimens will be collected at days 0, 10 and 70 to assay for markers of inflammation and microbial and metabolic profiling. For those not able to, or who refuse in-person visits, the investigators will allow a virtual encounter and shipment of the study agent. If not able to come for in person visits, blood draws may be omitted and shipment of urine and stool specimens will be allowed. Sample collection containers will also be provided as needed for sample transport to the participants next scheduled follow-up visit.

The data set utilized for all initial baseline feature and demographic reporting will be the Intention to Treat Analysis Dataset, which will be comprised of all randomized participants. The primary dataset will be a Modified Intention to Treat Analysis Dataset for all endpoints, comprised of all participants who took at least one dose of study intervention (placebo or treatment), regardless of completeness of follow-up outcome data. The Safety Analysis Dataset will be all participants who took at least one dose of study intervention. The Per Protocol Analysis Dataset will be those patients who took at least 9 doses of study intervention for 9 days of the treatment period (10 days). Analysis will utilize ANOVA unless statistically significant differences in the distribution of baseline characteristics or features of non-normality are detected and relevant, at which point contingency utilization of ANCOVA, logistic regression, or other approaches as appropriate will be implemented. Treatment group level rates will be presented as incidence risk ratios relative to the control (placebo) group with 95% confidence intervals.

Safety endpoints will be evaluated on an individual AE by AE event via the DSMB and utilizing summary statistics during treatment and through duration of follow up. Adverse events will be presented by System Organ Class and will include information on start and stop date, severity, projected relationship, expectedness, and outcome and duration (the latter two after the event is considered to have concluded).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years and older.
4. Admitted to UVA hospital, or seen as an outpatient, or seen at Carilion hospital.
5. Presence of diarrhea*
6. Episode of C. difficile infection, non-severe or severe uncomplicated.
7. Within 120 hours of receiving standard therapy (oral vancomycin or fidaoxmicin).
8. Must be able to provide informed consent in person or electronically, or if not able to have a LAR to provide consent, in person or remotely via virtual or electronic means.

Exclusion Criteria:

1. At enrollment, presence of any of the following:

   1. Hypotension or shock
   2. Megacolon or moderate to severe ileus
   3. Acute abdomen
   4. Admission to intensive care unit
2. Inability to tolerate oral or enteral medication
3. Presence of other known infectious etiology of diarrhea
4. COVID-19 co-infection at the time of CDI diagnosis.
5. Absolute neutrophil count <500 mcl
6. Within 100 days of hematologic or solid organ transplant

   • Inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis) or other etiology of non-infectious diarrhea. For patients with history of IBD, allow enrollment if disease is well-controlled and stable (not in flare).
7. Enrollment in another investigational drug trial
8. Current use of alternative treatment for CDI (e.g. antibiotics other than vancomycin or fidaxomicin; IVIg; fecal transplant).
9. On probiotics and not willing to discontinue.
10. Cirrhosis or in participants with ALT > 3X normal
11. End stage renal disease, unless on dialysis(HD or PD) or creatinine clearance or estimated GFR of <30mL/min even after adequate hydration
12. Life expectancy of < 6 months.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrent CDI. | Within 60 days post-treatment
  Documented C difficile infection defined by presence of recurrent diarrhea with stool positive for C difficile assay necessitating treatment with anti-C. difficile antibiotic.

SECONDARY OUTCOMES:
Number of participants who died post-study treatment | Until 60 days post-treatment
  Documentation of death from any cause occurring during study treatment and 60 days after study treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UVA Health Systems, Charlottesville, Virginia
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication
Access Criteria: To be determined later.

REFERENCES:
- [Derived] Warren CA, Shin JH, Bansal EN, Costa DVDS, Wang XQ, Wu M, Swann JR, Behm BW, Targonski PV, Archbald-Pannone L. Alanyl-glutamine supplementation for Clostridioides difficile infection treatment (ACT): a double-blind randomised controlled trial study protocol. BMJ Open. 2023 Jul 19;13(7):e075721. doi: 10.1136/bmjopen-2023-075721. PMID 37474181